CLINICAL TRIAL: NCT00978367
Title: A Double Blind, Placebo (Vehicle) and Standard Care Controlled, Randomised Study to Investigate the Clinical Safety and Toleration (Including Systemic Pharmacokinetics), Wound Healing and Anti-scarring Potential of Two Applications of Intradermal RN1001 in Healthy Male Subjects.
Brief Title: Investigation of the Safety, Dosing Frequency and Anti-Scarring Potential of Two Concentrations of Intradermal Avotermin (Juvista)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: John Hutchison, Medical Director, Renovo Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RN1001-319-1003
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Cicatrix; Wound Healing; Re-epithelialization
Keywords: Cicatrix; Scar; Avotermin; Juvista; RN1001; TGF beta 3
MeSH Terms: conditions — Cicatrix | interventions — TGFB3 protein, human; Transforming Growth Factor beta3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug, intradermal avotermin (Juvista) (Experimental)
  Interventions: Drug: Avotermin
- Placebo (vehicle) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avotermin — 5 ng or 50 ng/100 ul avotermin applied by intradermal injection to one of two 3 mm punch biopsies on each arm just prior to surgery (on day 0) and again on day 5 just prior to excision of the wound with a 5 mm surgical ellipse
  Other Names: Juvista; RN1001; TGF beta 3
  Arms: Drug, intradermal avotermin (Juvista)
Drug: Avotermin — 5 ng or 50 ng/100 ul avotermin applied by intradermal injection to one of two 3 mm punch biopsies on each arm just prior to surgery (on day 0) and again on days 1 and 2. Dosing is repeated on day 5 (just prior to excision of the wound with a 5 mm surgical ellipse), 6 and 7.
  Other Names: Juvista; RN1001; TGF beta 3
  Arms: Drug, intradermal avotermin (Juvista)
Drug: Avotermin — 5 ng or 50 ng/100 ul avotermin applied by intradermal injection to one of two 3 mm punch biopsies on each arm just prior to surgery (on day 0) and again on days 1, 2, 3 and 4. Dosing is repeated on day 5 (just prior to excision of the wound with a 5 mm surgical ellipse), 6, 7, 8 and 9.
  Other Names: Juvista; RN1001; TGF beta 3
  Arms: Drug, intradermal avotermin (Juvista)
Drug: Placebo — Placebo applied by intradermal injection to one of two 3 mm punch biopsies on each arm just prior to surgery (on day 0) and again on day 5 just prior to excision of the wound with a 5 mm surgical ellipse
  Arms: Placebo (vehicle)
Drug: Placebo — Placebo applied by intradermal injection to one of two 3 mm punch biopsies on each arm just prior to surgery (on day 0) and again on days 1 and 2. Dosing is repeated on day 5 (just prior to excision of the wound with a 5 mm surgical ellipse), 6 and 7.
  Arms: Placebo (vehicle)
Drug: Placebo — Placebo applied by intradermal injection to one of two 3 mm punch biopsies on each arm just prior to surgery (on day 0) and again on days 1, 2, 3 and 4. Dosing is repeated on day 5 (just prior to excision of the wound with a 5 mm surgical ellipse), 6, 7, 8 and 9.
  Arms: Placebo (vehicle)

SUMMARY:
The purpose of this study is to investigate the dosing frequency, wound healing (re-epithelialisation) and anti-scarring effects of one, three and five applications of two concentrations of intradermal RN1001 in healthy male subjects.

DETAILED DESCRIPTION:
Subjects were randomised into two cohorts, to receive either 5 ng avotermin doses or 50 ng doses, with a minimum of 21 subjects per cohort. Within each cohort subjects were randomised into one of three dosing groups (7 subjects per group).

Subjects were to receive four 3 mm punch biopsies, two on the upper-inner aspect of each arm. One treatment was randomly allocated to one biopsy on one arm, with the opposite biopsy on the other arm set to receive the same treatment. The other treatment was administered to the other two biopsies (one on each arm. This allowed for control of possible positional effects on healing.

Three subjects per group received intradermal avotermin to one of the biopsies on each arm and intradermal placebo to the other biopsies. A different three subjects received intradermal avotermin to one of the biopsies on each arm and standard care only to the other biopsies. The final subject per group received intradermal placebo to one of the biopsies on each arm and standard care only to the other biopsy.

On day 0 biopsy sites were marked on both arms and following local anaesthesia avotermin, placebo or nothing was injected intradermally into the allocated sites. Subjects in dosing frequency group 1 (DFG 1) were dosed only once (day 0), subjects in DFG 2 were dosed three times (day 0, 1 and 2) and subjects in DFG 3 were dosed five times (day 0, 1, 2, 3 and 4).

On Day 5, all subjects had their punch biopsy wounds on one arm only re-dosed as per Day 0 and then excised with a 5 mm surgical ellipse. Subjects in DFG2 and DFG3 received further re-dosing on their excised punch biopsies as before, i.e. three doses for DFG2 and five doses for DFG3.

Subjects returned for a first follow-up at day 14 and then at months 2, 4 and 6 to examine for anti-scarring effects. At month 6 all scars were excised for histological examination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-Caribbean, male subjects aged 18-45 years inclusive
* Weight between 60-150 kg and a BMI within the permitted range for their height using Quetelet's index (15-45 kg/m(squared)) (weight (kg)/height (squared)(m))
* Subjects who have a previous history of surgery or minor injury and who have not developed any evidence of hypertrophic or keloid scar formation

Exclusion Criteria:

* Subjects who have a history or evidence of hypertrophic or keloid scarring
* Subjects with tattoos or previous scars in the area to be biopsied
* Subjects who have evidence of any past or present clinically significant disease, particularly coagulation disorders

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2002-02; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
To determine the dosing frequency of various concentrations of intradermal avotermin (Juvista) for the improvement of early wound healing and re-epithelialisation, as determined by measuring total wound diameter | Day 5 post surgery

SECONDARY OUTCOMES:
To determine the safety and toleration of various concentrations of avotermin (Juvista) applied by intradermal injection at various timepoints | Days 0-14 post-wounding
To determine the systemic exposure of various concentrations of avotermin (Juvista) applied by intradermal injection at various timepoints | Days 0-14 post-wounding
To determine the gross and histological endpoints (re-epithelialisation and wound healing) of various concentrations of avotermin (Juvista) applied by intradermal injection at various dosing frequencies | 0-6 months post-wounding
To determine the anti-scarring potential of two doses of avotermin (Juvista) when applied by intradermal injection at various dosing frequencies | Day 5 and 6 months post-wounding

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Davies, Principal Investigator — Renovo; Jonathan Duncan, Principal Investigator — Renovo
Locations (1):
- Renovo Ltd, Manchester, United Kingdom